CLINICAL TRIAL: NCT02750072
Title: INfrapatellar Versus SUprapatellar Reamed Intramedullary Nailing for Fractures of the Tibia
Acronym: INSURT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraser Orthopaedic Research Society (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FHREB #: 2016-029
Record Dates: First submitted 2016-04-18; First posted 2016-04-25 (Estimated); Last update posted 2024-01-30 (Actual); Status verified 2023-09

CONDITIONS: Tibial Fractures; Anterior Knee Pain Syndrome
MeSH Terms: conditions — Tibial Fractures; Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Infrapatellar approach (Active Comparator): Infrapatellar approach using the surgeon's incision of choice (i.e., patellar tendon split, tendon retraction medial, tendon retraction lateral).
  Interventions: Procedure: Infrapatellar Approach
- Semi-extended suprapatellar approach (Experimental): Semi-extended suprapatellar approach using quadriceps split combined with purpose designed suprapatellar percutaneous instrumentation (patellofemoral protection sleeve).
  Interventions: Procedure: Suprapatellar Approach

INTERVENTIONS:
Procedure: Infrapatellar Approach — Infrapatellar approach using the surgeon's incision of choice (i.e. patellar tendon split, tendon retraction medial, tendon retraction lateral)
  Arms: Infrapatellar approach
Procedure: Suprapatellar Approach — Semi-extended suprapatellar approach using quadriceps split combined with purpose designed percutaneous instrumentation
  Arms: Semi-extended suprapatellar approach

SUMMARY:
This study will investigate the incidence and severity of anterior knee pain comparing two different approaches to tibial nail fixation; Infrapatellar versus percutaneous semi-extended suprapatellar incisions. Half the patients will be randomized to the gold standard infrapatellar approach with the other half being randomized to treatment with the percutaneous semi-extended suprapatellar approach.

DETAILED DESCRIPTION:
There are a number of ways to approach the tibial canal when using an intramedullary nail for fracture fixation.

The gold standard is the infrapatellar approach (below the knee cap). This approach has the patient positioned with the knee flexed at 90 degrees or greater on the operating table. However, there are challenges with this approach, including imaging, placement of supplemental fixation, conversion to open reduction when necessary and malunion with apex anterior angulation for proximal tibial fractures. The positioning of the patient causes tension on the structures and soft tissues around the knee which can hinder the placement of the nail and can cause damage to the soft tissues that can result in significant long-term anterior knee pain for many patients.

The semi-extended suprapatellar approach has the patient positioned in approximately 15-20 degrees of flexion, putting less tension on the structures and soft tissues about the knee and enables the surgeon to insert the nail in an optimal position with relative ease.

ELIGIBILITY:
Inclusion Criteria:

* all extra-articular tibial fractures
* simple distal tibial intra-articular fractures amenable to IMN
* open and closed fractures
* bilateral tibiae
* willing and able to consent, follow protocol and attend follow-up visits
* able to read and understand English or have interpreter available

Exclusion Criteria:

* patients with contralateral femur and/or hip fracture requiring retrograde IMN
* patients with contralateral knee injuries that would impair their ability to kneel during the follow-up period
* associated knee injury
* previous symptomatic knee pathology
* ipsilateral injuries to the same limb that would interfere with rehab or outcome
* neurovascular injuries at the level of the knee requiring surgery
* open or closed fractures > 14 days (times of injury to OR)
* non unions
* pathologic fractures
* periprosthetic fractures
* spinal injury
* non-ambulatory patients
* incarceration
* limited life expectancy due to significant medical co-morbidities or medical contra-indication to surgery (pregnancy)
* likely problems, in the judgment of the investigators, with maintaining follow-up

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-10-12 (Actual)

PRIMARY OUTCOMES:
VAS (visual analog scale) for pain on kneeling/ability to knee | 12 months post treatment
  Participants assessment of their degree/level of pain on kneeling after performing the AKT (Aberdeen Kneeling Weight-Distribution Test) on a 10 cm visual analog scale

SECONDARY OUTCOMES:
AKT (Aberdeen Kneeling Weight-Distribution Test) | 4, 6, 12 and 24 months post treatment
  The AKT involves kneeling on two separate calibrated scales for up to 60 seconds with the patient blinded to the readings. At 15-second intervals the weight distribution, measured in kg, between the two knees is documented.
AST (Aberdeen Standing Weight-Distribution Test) | 4, 6, 12 and 24 months post treatment
  The AST involves the patient standing on two separate calibrated scales (one foot on each scale) and the weight in kg recorded with the patient blinded to the readings.
VAS (Visual Analog Scale) at rest, with walking and descending stairs | 4, 6, 12 and 24 months post treatment
  Participants overall assessment of their pain at rest, with walking and descending stairs over the past week on a 10 cm visual analog scale
Lysholm Knee Scoring Scale | 4, 6, 12 and 24 months post treatment
  Used to evaluate outcomes of knee ligament surgery using 8-items commonly affecting patients with anterior knee pain: Limp, support, locking, instability, pain, swelling, stair climbing and squatting.
PKPM (Photographic knee pain map) | 4, 6,12 and 24 months post treatment
  Used to determine the precise location of the knee pain, as indicated and localized by the participant.
EQ-5D Health Related Quality of Life Outcome Measure | 4, 6,12 and 24 months post treatment
  5 dimensions: Mobility: self-care, usual activities, pain/discomfort and anxiety/depression
WPAI:SHP (Work Productivity and Activity Impairment: Specific Health Problem | 4, 6, 12 and 24 months post treatment
  A questionnaire pertaining to the effect of the participants tibial fracture on their ability to work and perform regular activities.
Radiographic outcome | Intra-operatively and 4, 6,12 and 24 months post treatment
  Blinded independent reviewer will adjudicate alignment, nail position and determination of union at one year, as well as change of position of the nail.

CONTACTS AND LOCATIONS:
Overall Officials: Darius G Viskontas, MD, FRCSC, Principal Investigator — Royal Columbian Hospital / Fraser Health Authority; Trevor B Stone, MD, FRCSC, Principal Investigator — Royal Columbian Hospital / Fraser Health Authority; Alan Johnstone, Professor, Principal Investigator — Aberdeen Royal Infirmary
Locations (6):
- Canada (5):
  - University of Alberta Hospital, Edmonton, Alberta
  - Royal Columbian Hospital / Fraser Health Authority, New Westminster, British Columbia
  - Hamilton Health Sciences, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karachalios T, Babis G, Tsarouchas J, Sapkas G, Pantazopoulos T. The clinical performance of a small diameter tibial nailing system with a mechanical distal aiming device. Injury. 2000 Jul;31(6):451-9. doi: 10.1016/s0020-1383(00)00024-3. PMID 10831746
- [Background] Toivanen JA, Vaisto O, Kannus P, Latvala K, Honkonen SE, Jarvinen MJ. Anterior knee pain after intramedullary nailing of fractures of the tibial shaft. A prospective, randomized study comparing two different nail-insertion techniques. J Bone Joint Surg Am. 2002 Apr;84(4):580-5. doi: 10.2106/00004623-200204000-00011. PMID 11940618
- [Background] Katsoulis E, Court-Brown C, Giannoudis PV. Incidence and aetiology of anterior knee pain after intramedullary nailing of the femur and tibia. J Bone Joint Surg Br. 2006 May;88(5):576-80. doi: 10.1302/0301-620X.88B5.16875. No abstract available. PMID 16645100
- [Background] Weninger P, Schultz A, Traxler H, Firbas W, Hertz H. Anatomical assessment of the Hoffa fat pad during insertion of a tibial intramedullary nail--comparison of three surgical approaches. J Trauma. 2009 Apr;66(4):1140-5. doi: 10.1097/TA.0b013e318169cd4d. PMID 19359927
- [Background] Koval KJ, Clapper MF, Brumback RJ, Ellison PS Jr, Poka A, Bathon GH, Burgess AR. Complications of reamed intramedullary nailing of the tibia. J Orthop Trauma. 1991;5(2):184-9. doi: 10.1097/00005131-199105020-00011. PMID 1650401
- [Background] Ryan SP, Steen B, Tornetta P 3rd. Semi-extended nailing of metaphyseal tibia fractures: alignment and incidence of postoperative knee pain. J Orthop Trauma. 2014 May;28(5):263-9. doi: 10.1097/BOT.0000000000000083. PMID 24751605
- [Background] Jones M, Parry M, Whitehouse M, Mitchell S. Radiologic outcome and patient-reported function after intramedullary nailing: a comparison of the retropatellar and infrapatellar approach. J Orthop Trauma. 2014 May;28(5):256-62. doi: 10.1097/BOT.0000000000000070. PMID 24464093
- [Background] Vaisto O, Toivanen J, Paakkala T, Jarvela T, Kannus P, Jarvinen M. Anterior knee pain after intramedullary nailing of a tibial shaft fracture: an ultrasound study of the patellar tendons of 36 patients. J Orthop Trauma. 2005 May-Jun;19(5):311-6. PMID 15891539
- [Background] Leliveld MS, Verhofstad MH. Injury to the infrapatellar branch of the saphenous nerve, a possible cause for anterior knee pain after tibial nailing? Injury. 2012 Jun;43(6):779-83. doi: 10.1016/j.injury.2011.09.002. Epub 2011 Oct 1. PMID 21962297
- [Background] Cartwright-Terry M, Snow M, Nalwad H. The severity and prediction of anterior knee pain post tibial nail insertion. J Orthop Trauma. 2007 Jul;21(6):381-5. doi: 10.1097/BOT.0b013e3180caa138. PMID 17620996
- [Background] Vaisto O, Toivanen J, Kannus P, Jarvinen M. Anterior knee pain after intramedullary nailing of fractures of the tibial shaft: an eight-year follow-up of a prospective, randomized study comparing two different nail-insertion techniques. J Trauma. 2008 Jun;64(6):1511-6. doi: 10.1097/TA.0b013e318031cd27. PMID 18545115
- [Background] Tornetta P 3rd, Collins E. Semiextended position of intramedullary nailing of the proximal tibia. Clin Orthop Relat Res. 1996 Jul;(328):185-9. doi: 10.1097/00003086-199607000-00029. PMID 8653954
- [Background] Sanders RW, DiPasquale TG, Jordan CJ, Arrington JA, Sagi HC. Semiextended intramedullary nailing of the tibia using a suprapatellar approach: radiographic results and clinical outcomes at a minimum of 12 months follow-up. J Orthop Trauma. 2014 Aug;28 Suppl 8:S29-39. doi: 10.1097/01.bot.0000452787.80923.ee. PMID 25046413
- [Background] Morandi M, Banka T, Gaiarsa GP, Guthrie ST, Khalil J, Hoegler J, Lindeque BG. Intramedullary nailing of tibial fractures: review of surgical techniques and description of a percutaneous lateral suprapatellar approach. Orthopedics. 2010 Mar;33(3):172-9. doi: 10.3928/01477447-20100129-22. No abstract available. PMID 20205366
- [Background] Kubiak EN, Widmer BJ, Horwitz DS. Extra-articular technique for semiextended tibial nailing. J Orthop Trauma. 2010 Nov;24(11):704-8. doi: 10.1097/BOT.0b013e3181d5d9f4. PMID 20881632
- [Background] Court-Brown CM, Gustilo T, Shaw AD. Knee pain after intramedullary tibial nailing: its incidence, etiology, and outcome. J Orthop Trauma. 1997 Feb-Mar;11(2):103-5. doi: 10.1097/00005131-199702000-00006. PMID 9057144
- [Background] Song SY, Chang HG, Byun JC, Kim TY. Anterior knee pain after tibial intramedullary nailing using a medial paratendinous approach. J Orthop Trauma. 2012 Mar;26(3):172-7. doi: 10.1097/BOT.0b013e3182217fe6. PMID 22068208
- [Background] Courtney PM, Boniello A, Donegan D, Ahn J, Mehta S. Functional Knee Outcomes in Infrapatellar and Suprapatellar Tibial Nailing: Does Approach Matter? Am J Orthop (Belle Mead NJ). 2015 Dec;44(12):E513-6. PMID 26665254
- [Background] Garratt AM, Brealey S, Gillespie WJ; DAMASK Trial Team. Patient-assessed health instruments for the knee: a structured review. Rheumatology (Oxford). 2004 Nov;43(11):1414-23. doi: 10.1093/rheumatology/keh362. Epub 2004 Aug 17. PMID 15316121
- [Background] Lysholm J, Gillquist J. Evaluation of knee ligament surgery results with special emphasis on use of a scoring scale. Am J Sports Med. 1982 May-Jun;10(3):150-4. doi: 10.1177/036354658201000306. PMID 6896798
- [Background] Tegner Y, Lysholm J. Rating systems in the evaluation of knee ligament injuries. Clin Orthop Relat Res. 1985 Sep;(198):43-9. PMID 4028566
- [Background] Elson DW, Jones S, Caplan N, Stewart S, St Clair Gibson A, Kader DF. The photographic knee pain map: locating knee pain with an instrument developed for diagnostic, communication and research purposes. Knee. 2011 Dec;18(6):417-23. doi: 10.1016/j.knee.2010.08.012. Epub 2010 Sep 17. PMID 20850976
- [Background] Leighton RK, Trask K. The Canadian Orthopaedic Trauma Society: a model for success in orthopaedic research. Injury. 2009 Nov;40(11):1131-6. doi: 10.1016/j.injury.2008.11.021. Epub 2009 Apr 21. PMID 19386310
- [Background] Crossley KM, Bennell KL, Cowan SM, Green S. Analysis of outcome measures for persons with patellofemoral pain: which are reliable and valid? Arch Phys Med Rehabil. 2004 May;85(5):815-22. doi: 10.1016/s0003-9993(03)00613-0. PMID 15129407
- [Background] Mills K, Blanch P, Vicenzino B. Identifying clinically meaningful tools for measuring comfort perception of footwear. Med Sci Sports Exerc. 2010 Oct;42(10):1966-71. doi: 10.1249/MSS.0b013e3181dbacc8. PMID 20216463
- [Background] Hinman RS, McCrory P, Pirotta M, Relf I, Forbes A, Crossley KM, Williamson E, Kyriakides M, Novy K, Metcalf BR, Harris A, Reddy P, Conaghan PG, Bennell KL. Acupuncture for chronic knee pain: a randomized clinical trial. JAMA. 2014 Oct 1;312(13):1313-22. doi: 10.1001/jama.2014.12660. PMID 25268438